CLINICAL TRIAL: NCT07020078
Title: Salivary Redox Biomarkers in Relation to Oral Health Condition Among a Group of Ionizing Radiation Field Workers
Brief Title: Oral Health Condition Among a Group of Ionizing Radiation Field Workers
Status: Not yet recruiting | Type: Observational
Sponsor: Al-Mustansiriyah University (Other)
Responsible Party: Principal Investigator, Jihan munther hussien, Master student, Al-Mustansiriyah University
Other Study IDs: MustansiriyahU
Record Dates: First submitted 2025-05-04; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-04

CONDITIONS: Salivary Redox Biomarkers and Oral Health

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Salivary redox biomarkers — Salivary redox biomarkers

SUMMARY:
The goal of this study is to test the effect of ionizing radiation on salivary Redox status among a group of ionizing radiation workers by measuring salivary biomarkers(malondialdehyde,8_hydroxy_deoxyguanosine and catalase) and measuring oral health condition by plaque index.

90 male subjects will be enrolled in this study between 30_40 years old worked in Baghdad teaching hospital ,30 subjects exposed from computed tomography department ,30 subjects exposed from x_ray department and 30 subjects unexposed from laboratory department in the same hospitals.

The method of the study is taking unstimulated saliva sample from the subjects and oral health measure.

ELIGIBILITY:
Inclusion Criteria:

* male, 30_40 years ,no history of systemic disease, no medical treatment taken at least 3 months before sampling and the subjects are exposed to radiation 5_ 10 years

Exclusion Criteria:

* subjects with medical history , subjects are taken medications during last 3 months , the subjects are exposed to radiation less than 5 years or more than 10 years

Ages: 30 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Male workers in radiation field from 30_40 years old who exposed to radiation for 5_10 years and compare them with male workers in laboratory at age 30_40 years
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-06-25 (Estimated); Primary Completion 2025-07-25 (Estimated); Study Completion 2025-08-25 (Estimated)

PRIMARY OUTCOMES:
oral health status | Baseline: the subjects must be fasting. up to two hours saliva collection
  Changes in the clinical periodontal parameter (Plaque index ) To determine the patients' plaque index, their dental plaque thickness was evaluated by probing the mesial, distal, buccal, and palatal surfaces of all teeth using a Williams periodontal probe. The individual's plaque index was determined by summing the values obtained for each tooth and calculating the averages.Silness & Löe (Silness & Löe,1964) reference values were taken as a basis The Plaque Index (PI) scores each site on a 0 to 3 scale Score 0 : No plaque is in the area adjacent to the gingiva. Score 1: There is a plaque in the form of a thin film on the gingival margin. Score 2: There is a visible plaque in the gingival pocket and gingival margin. Score 3: There is a dense plaque in the gingival pocket and on the gingival margin.

SECONDARY OUTCOMES:
Salivary Malondialdehyde biomarker | Baseline:saliva collection for malondialdehyde . up to two hours fasting for all subjects.
  Measure salivary malondialdehyde biomarker for all 90 subjects (computed tomography,x_ray and laboratory group) to see if the ionizing radiation effect on salivary Redox status in relation to oral health condition for workers in radiation field
Salivary 8_ hydroxy_deoxyguanosine biomarker | Baseline:saliva collection for 8_hydroxy_deoxyguanosine .up to two hours fasting for all subjects.
  Measure salivary 8_hydroxy_deoxyguanosine biomarker for all 90 subjects (computed tomography,x_ray and laboratory group) to see if the ionizing radiation effect on salivary Redox status in relation to oral health condition for workers in radiation field
Salivary catalase biomarker | Baseline:saliva collection for catalase . up to two hours fasting for all subjects.
  Measure salivary catalase biomarker for all 90 subjects (computed tomography,x_ray and laboratory group) to see if the ionizing radiation effect on salivary Redox status in relation to oral health condition for workers in radiation field

IPD SHARING:
Plan to Share IPD: No